CLINICAL TRIAL: NCT05338242
Title: Environmental Exposures of the Northern Arapaho Tribe: An Exploratory Study
Brief Title: Monitoring Environmental Exposures and Behavioral Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Darrah Sleeth, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21NArapaho; R21ES032137 (NIH)
Record Dates: First submitted 2022-04-13; First posted 2022-04-21 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Risk Reduction; Environmental Exposure; Risk Behavior, Health
MeSH Terms: conditions — Risk Reduction Behavior; Health Risk Behaviors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real-Time Feedback (Experimental): Participants will receive real-time exposure monitors that continuously display real-time air concentration information and a color-coded designation for the current risk level.
  Interventions: Device: Real-Time Exposure Feedback
- No Feedback (No Intervention): Participants will have exposure levels monitored by the same device, but it will only display the date/time and will not provide real-time feedback.

INTERVENTIONS:
Device: Real-Time Exposure Feedback — Participants will receive real-time exposure monitors that continuously display real-time air concentration information and a color-coded designation for the current risk level.
  Arms: Real-Time Feedback

SUMMARY:
The goal of this study is to examine what effect real-time feedback on particulate matter (PM) air pollution levels has on risk recognition and behavior. The hypothesis is that real-time exposure feedback will change perceptions of risk and increase behaviors that avoid exposure to environmental risks. At least one representative household member in participating households will complete a questionnaire to fully understand environmental concerns, risk perceptions, and related behaviors. Half of the households will have PM monitors that continuously display real-time concentrations and an indication of the hazard level. The other participants will have the same device but it will only display the date and time. All participants will then be surveyed again: (a) immediately after sampling is complete (i.e., when the devices are removed from the home), (b) after 3 months and, (c) after 6 months. The goal of repeated surveys is to determine changing understanding of risks, how participating in research and/or receiving real-time exposure data may have changed participant behavior, and what concerns they continue to have. The questionnaire will include questions with categorical and/or quantitative answers (e.g., frequency of specific behaviors) so that changes in risk perception and behavior can be effectively analyzed.

ELIGIBILITY:
Participants must live in a household where at least one adult is a member of the N. Arapaho tribe who is a Primary Participant in the related exposure assessment study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Behaviors Related to Reduction in Exposure | At removal of device
  Outcomes will be measured as a change in how often (frequency) behaviors related to reduction in exposure occur
Behaviors Related to Reduction in Exposure | 3 months after removal of device
  Outcomes will be measured as a change in how often (frequency) behaviors related to reduction in exposure occur
Behaviors Related to Reduction in Exposure | 6 months after removal of device
  Outcomes will be measured as a change in how often (frequency) behaviors related to reduction in exposure occur

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No